CLINICAL TRIAL: NCT04989335
Title: An Open-label, Phase II, Two-stage, Study of Bisantrene(Xantrene) in Combination With Fludarabine and Clofarabine as Salvage Therapy for Adult Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Bisantrene Combination for Resistant AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Race Oncology Ltd (Industry)
Responsible Party: Principal Investigator, Prof Arnon Nagler, Director Hematology Division, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC-002
Record Dates: First submitted 2021-07-07; First posted 2021-08-04 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Myelogenous Leukemia, Acute
Keywords: AML, Resistance relapsing ,Anti Leukemic effect , Bisantrene
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — bisantrene; fludarabine; Clofarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bisantrene combined with Fludarabine and Clofarabine (Experimental): Bisantrene 250 mg at final concentration of 0.5 mg/mL will be administrated by intravenous (IV) infusion, delivered by a controlled-rate programmable pump via a central line over 2 hours.
  Fludarabine (generic) and Clofarabine (generic) are commercially available as injection for intravenous infusion.
  The treatment regimen will comprise daily IV infusion of Fludarabine (Flu), Clofarabine (Clo) and Bisantrene (Xan) administered via central venous line and controlled-rate infusion pump with a 1-hour break between each agent infusion, amounting to a total of 6 hours for each daily FluCloXan treatment in the following sequence:
  * First, infusion over 60 minutes of Fludarabine (Flu) at 10 mg/m2
  * Followed by infusion of Clofarabine (Clo) at 30 mg/m2 over 60 minutes
  * Followed by infusion of Bisantrene (Xan) at 250 mg/m2 over 2 hours.
  Interventions: Drug: Bisantrene; Drug: Fludarabine; Drug: Clofarabine

INTERVENTIONS:
Drug: Bisantrene — Combined escalated dose chemotherapy
Drug: Fludarabine — Combined escalated dose chemotherapy
Drug: Clofarabine — Combined escalated dose chemotherapy

SUMMARY:
An Open-label, Phase II, Two-stage, Study of Xantrene® (Bisantrene) in combination with Fludarabine and Clofarabine as Salvage Therapy for Adult Patients with Relapsed or Refractory Acute Myeloid Leukemia (AML) Lead-in stage: up to 12 (up to 2 cohorts in a 3+3 dose escalation design) Efficacy stage: up to 17 (Simon 2-stage design 9+8)

Study Objectives:

* Confirm safety and tolerability of the combination regimen
* Time to response with combination treatment
* Overall survival

The treatment regimen will comprise daily IV infusion of Fludarabine (Flu), Clofarabine (Clo) and Bisantrene (Xan) administered via central venous line and controlled-rate infusion pump with a 1-hour break between each agent infusion, amounting to a total of 6 hours for each daily FluCloXan treatment in the following sequence:

* First, infusion over 60 minutes of Fludarabine (Flu) at 10 mg/m2
* Followed by infusion of Clofarabine (Clo) at 30 mg/m2 over 60 minutes
* Followed by infusion of Bisantrene (Xan) at 250 mg/m2 over 2 hours. One cycle will comprise daily IV infusion of the combination treatment course for 4 or 5 consecutive days and rest period to between Day 30 and Day 42, based on patient performance and disease status.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent and privacy language as per national regulations.
2. Age 18 -65 (inclusive) years
3. Diagnosis of AML by World Health Organization (WHO) classification (WHO, 2016) and have received at least one line of therapy prior to enrollment into this study.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.0
5. Life expectancy ≥ 3 months.
6. Adequate organ function as evidenced by serum total bilirubin ≤ 2.0 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤4 × the upper limit of normal (ULN), serum albumin >2.8 g/dL, serum creatinine ≤2 mg/dL.
7. Cardiac ejection fraction ≥50%, assessed by 2-Dimensional echocardiogram.
8. Pulmonary function ≥50% assessed by diffusing capacity for carbon monoxide (DLCO), and any clinically significant decrease in DLCO must not be caused by infection.
9. Negative for serum markers for HIV, Hepatitis -B, -C, and HTLV-1
10. Clinically significant non-hematologic toxicity after prior chemotherapy has recovered to Grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
11. Females must be surgically or biologically sterile or postmenopausal (amenorrhoeic for at least 12 months) or if of childbearing potential, must have a negative urine or serum pregnancy test within 14 days before study entry, and must agree to use an adequate method of contraception, i.e. barrier method, during the study until 30 days after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception, i.e. barrier method, during the study until 30 days after the last treatment.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APML, APL) M3 subtype of AML.
2. Other active malignancy (including other hematologic malignancies) or other malignancy within the last 12 months except non-melanoma skin cancer or cervical intraepithelial neoplasia.
3. Prior or current therapy:

   1. Hydroxyurea or other oral medications to reduce blast count within 72 hours before the first dose of study drug
   2. Treatment with an investigational agent within 14 days before the first dose of study drug, or not recovered from all acute effects of previous investigational therapy
   3. Last treatment was with a drug of long elimination half-life (e.g. enasidenib), as such a wash out period 5x elimination half-life is necessary prior to enrollment
4. For patients who have undergone hematopoietic stem cell transplantation (HSCT), procedure-related medications (e.g. immunosuppressive therapy) administered within 2 weeks prior to first dose of study drug.
5. Any medical, psychological, or social condition that may interfere with study participation or compliance or may compromise the patient's safety in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The recommended Phase 2 dose (RP2D) , assessed by the number of treatment days of FluCloXan | 12 months
The maximum tolerated dose (MTD) of Bisantre in mg per day | 12 months
  To evaluate safety and tolerability
The overall response rate (ORR) | between Day 30 to Day 42.
  Overall Response Rate (ORR) defined as the proportion of patients with complete remission (CR) and complete remission with incomplete blood count recovery (CRi) between Day 30 to Day 42.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 12 months
  Confirm safety and tolerability of the combination regimen.
Time of respons in months | 12 months
  Number of months for each patient with no evidence of diseases.
Overall survival | 12 months
  Median surviving months for each patients.

OTHER OUTCOMES:
MRD status | 12 months
  To determine the MRD status of patients post completion of FluCloXan. MRD will be asset in patients with defiant mutations by Polymerase Chain Techniques(PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel